CLINICAL TRIAL: NCT05072093
Title: Parrying the Pitfalls of PrEP: Preventing Premature PrEP Discontinuation and STIs Among MSM
Brief Title: Parrying the Pitfalls of PrEP: Project PEACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000608; 5R01MH123724-02 (NIH)
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: HIV; STI
Keywords: Prevention; Doxycycline; Apretude
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Doxycycline; cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All men in cohort: MSM (Experimental): Prospective cohort of MSM who are followed either in-person at the PRISM Health Research Clinic and/or virtually with remote study visits. Participants will have the option to switch prevention options at any point during the study by indicating their interest during monthly surveys or contacting study staff directly.
  Interventions: Behavioral: PrEP discontinuation intervention; Drug: Offering of on-demand oral PrEP; Drug: Offering of STI PEP; Drug: Injectable PrEP

INTERVENTIONS:
Behavioral: PrEP discontinuation intervention — Men taking daily oral PrEP (Truvada) will receive a monthly screener through the mobile app. If answers to screener questions indicate a participant is at risk for PrEP discontinuation, then a peer navigator will deliver a motivational interviewing intervention and a clinician will consult with the participant. These efforts are intended to avert PrEP discontinuation.
Drug: Offering of on-demand oral PrEP — For men who are not interested in daily oral PrEP or plan to discontinue daily oral PrEP, the investigators will offer on-demand oral PrEP (Truvada) which will allow them to take it immediately before/after a sexual encounter. It is hoped that this will serve as an alternative to daily oral PrEP use that is desirable for some people.
  Other Names: emtricitabine/tenofovir disoproxil, Truvada
Drug: Offering of STI PEP — All men in the cohort will be offered STI PEP (doxycycline) to use after condomless sex with the goal of averting STI diagnoses. At a dosage of 200 mg to be taken in a single dose ideally within 24 hours of possible exposure (e.g. condomless anal sex) and no later than 72 hours after exposure. Participants will be dispensed enough pills to allow for up to 3 weekly doses of 200mg doxycycline (i.e. 6 pills/week) for 3 months (the interval between STI testing visits).
  Other Names: doxycycline
Drug: Injectable PrEP — For men who are interested in injectable PrEP, they will be referred to local providers to access Apretude (Cabotegravir injection) every two months. In the study, their use of the medication will be monitored through monthly surveys during which they have the option to indicate interest in switching to oral PrEP.
  Other Names: Apretude, Cabotegravir

SUMMARY:
The study is a prospective cohort of young MSM who are followed for 2 years either in-person at the PRISM Health Research Clinic and/or virtually with telehealth study visits. Follow-up visits occur as frequently as every 3 months, or as appropriate to clinical needs of HIV PrEP or STI PEP. The investigators will enroll men who may decide to start or stop PrEP, change from daily oral PrEP to on-demand oral PrEP or from on-demand oral PrEP to daily PrEP, to start or stop STI PEP at any point in the study period, or injectable PrEP as an alternative to daily oral PrEP or on-demand oral PrEP. All men will be provided with the study's mobile smart phone app to support early identification of risks for PrEP discontinuation, to provide information about STI PEP and document usage patterns of on-demand oral PrEP and STI PEP, and to support easy linkage to support services for PrEP counseling and addressing concerns or questions about STI PEP and injectable PrEP.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) are disproportionately impacted by the U.S. HIV epidemic. Pre-exposure prophylaxis, or PrEP, is a relatively newer HIV prevention strategy that involves taking HIV antiviral medications either daily or on-demand to prevent HIV infection following high risk sexual activity. Both daily and on-demand PrEP have been shown to prevent infection if taken consistently and correctly. A prior research with this high-risk population in Atlanta, where it was offered daily PrEP to study participants, resulted in significant PrEP interest and initiation however high rates of PrEP discontinuation throughout the study were of great concern and, in some cases, led to HIV infection. Additionally, the study found high rates of bacterial sexually transmitted infection (STI) diagnoses both independent of, and concurrent with, higher PrEP use leading to concerns that condoms are not being used among MSM on PrEP.

The proposed work will expand upon the previous study with an intervention focus for MSM in Atlanta with aims of (1) preventing daily oral PrEP discontinuation; (2) offering on-demand oral PrEP as an alternative for MSM not interested in daily oral PrEP, (3) decreasing the incidence of bacterial STIs by offering STI post-exposure prophylaxis (PEP) which involves taking doxycycline immediately following high risk sexual behavior, 4) to start injectable PrEP as an alternative to daily oral PrEP or on-demand PrEP.

The study will involve a cohort of 200 MSM aged 18-45 in Atlanta who will be followed for two years. Participants will be recruited online from social media and dating websites, and in-person from different venues and events where MSM are known to attend. Men will take a short online eligibility screener either on a tablet, if recruited in-person, or on their own device if recruited online. Participants will be compensated for the various study activities (e.g., study visits, online behavioral surveys, weekly/monthly surveys).

If men screen eligible, they will be invited to a baseline study visit that will occur either in-person at the research clinic or virtually. Because of the ongoing COVID-19 pandemic, the plan is to offer participants the option of conducting study activities virtually or in-person. Consent will occur at the beginning of the baseline visit. Following the baseline visit, all participants will have two more study visits at months 12 and 24. At the three study visits, participants will be tested for HIV, STIs and drugs of abuse and take an online behavioral survey. Participants will also take an online behavioral survey at months 4, 7 and 19.

At all study visits, participants will discuss with the study counselor the various prevention options the study is offering-daily PrEP, on-demand PrEP, STI PEP or injectable PrEP as an alternative to daily oral PrEP or on-demand oral PrEP. If a participant elects to begin any of these, study staff will assist them in accessing oral PrEP from a community pharmacy and STI PEP (doxycycline) from the Emory Investigational Drug Service. Participants who start oral PrEP and/or STI PEP will take short weekly surveys for the first 2 weeks to monitor use and side effects. Following that 2-week period, daily oral PrEP users will get a monthly survey to try and detect warning signs of discontinuation so that the study can intervene to prevent that from happening. On-demand oral PrEP and STI PEP users will continue to get weekly surveys to monitor use and side effects. Oral PrEP and STI PEP users will have a 3-monthly visit-either in-person or virtually-to monitor their use and to test for HIV and STIs. Oral PrEP users will also have their kidney function monitored by creatinine testing. Participants electing to do their study activities virtually will be sent specimen collection kits so that they can self-collect specimens for all the required labs. They will mail back the specimens to the lab in a pre-paid postage mailer. Participants who elect injectable PrEP will be referred to local providers to access the medication; as part of our study, we will monitor their use through monthly surveys. Injectable PrEP Participants will have the option to switch prevention options at any point during the study by indicating their interest during monthly surveys or contacting study staff directly. Study clinicians will develop transition plan based on clinical indications.

All participants will be required to download the study app at the baseline visit and will be oriented to using it to retrieve study communication, surveys, lab results, etc. Additionally, the app will be used to schedule and conduct video conferencing sessions between participants and study clinicians/staff. If a participant reports warning signs of daily PrEP discontinuation, a peer navigator on staff will reach out through the app to try and schedule a counseling session that will use a motivational interviewing approach to support PrEP persistence.

The proposed work is of great significance for the field as novel approaches to preventing early discontinuation of PrEP are of utmost importance for preventing HIV transmission among MSM. If engaging with them frequently and assessing for warning signs of discontinuation is shown to be an effective strategy for intervening and preventing stoppage, then the implications for future interventions by community PrEP providers and clinicians is significant.

ELIGIBILITY:
Inclusion Criteria:

* Male at birth
* Self-identify as Cisgender Male
* Ages 18-45 years
* ≥1 male anal sex partner in the 12 months before the baseline interview
* Live in the Atlanta MSA
* Owns cell phone with data service
* Willing to download a health-related app to their cell phone as part of the research study
* Able to provide ≥ 2 means of contact
* Not currently enrolled in another HIV prevention clinical trial
* Confirmed HIV-negative at baseline visit

Exclusion Criteria:

* Female at birth
* Do not self-identify as Cisgender Male
* Individuals < 18 years of age or > 45 years of age
* HIV positive status
* No male anal sex partner in the 12 months before the baseline interview
* Does not own mobile phone with data service
* Not willing to download a health-related app to their cell phone as part of the research study
* Live outside the metro Atlanta MSA and/or planning to move from Atlanta area in the next 2 years
* Currently enrolled in an HIV prevention or treatment clinical trial
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males at birth are eligible for the study
Enrollment: 240 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Number of men who discontinue daily oral PrEP | 24 month post intervention
  MSM taking daily oral PrEP will complete monthly screener surveys delivered through study app to assess for PrEP stop intentions. After early identification, they will receive Motivational Interviewing (MI) to avoid discontinuation. Participants that discontinue PrEP will be measured.
Number of men who initiate on-demand oral PrEP | 24 month post intervention
  MSM who decline daily oral PrEP will be prescribed TDF/FTC fixed dose combination, 2 doses 2-24 hrs before sex and single dose 24 and 48 hours after first dose.
Number of men who initiate long-acting injectable PrEP | 24 month post intervention
  Number of men who are not interested in daily oral PrEP or on-demand oral PrEP will be offered Long-acting injectable PrEP through referral to outside providers.
Change in number of STI diagnoses from baseline at 12 and 24 months | Baseline, 12 and 24 months post intervention
  All men in cohort will be evaluated for STI diagnoses after 12 and 24 month post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sullivan, MD, Principal Investigator — Emory University
Locations (1):
- PRISM Research Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication will be shared, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following primary publication.
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.
  Proposals should be directed to pssulli@emory.edu. To gain access, data requestor will need to sign a data access agreement.

REFERENCES:
- [Derived] Aldredge A, Carter D, DeCree CA, Gardner EV, Herring GB, Kaabi O, Moges-Banks R, Valencia R, Kelley CF, Sullivan PS. Preventing Premature Pre-Exposure Prophylaxis Discontinuation and Sexually Transmitted Infections Among Men Who Have Sex With Men (Project PEACH): Protocol for a Prospective Cohort Study. JMIR Res Protoc. 2025 Apr 23;14:e56096. doi: 10.2196/56096. PMID 40267471

DOCUMENTS (1):
  • Informed Consent Form (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT05072093/ICF_000.pdf